CLINICAL TRIAL: NCT03870997
Title: Influenza Vaccination Digital Interventions for People Living With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidation Health (Industry)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EH-008
Record Dates: First submitted 2019-03-07; First posted 2019-03-12 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diabetes Digital Intervention (Experimental)
  Interventions: Behavioral: Diabetes Digital Intervention
- Generic Digital Intervention (Experimental)
  Interventions: Behavioral: Generic Digital Intervention
- No Influenza Vaccination Intervention (No Intervention)

INTERVENTIONS:
Behavioral: Diabetes Digital Intervention — The Diabetes Digital Intervention is a digital campaign that provides interactive ways (e.g., videos, infographics, quizzes) for individuals to learn about influenza and related complications, and the importance of influenza vaccination. It is tailored to people living with diabetes and highlights the importance of influenza vaccination for this specific patient population.
  Arms: Diabetes Digital Intervention
Behavioral: Generic Digital Intervention — The Generic Digital Intervention is a digital campaign that provides interactive ways (e.g., videos, infographics, quizzes) for individuals to learn about influenza and related complications, and the importance of influenza vaccination. It provides generic influenza vaccination interventions that can be applicable to any adult who should receive influenza vaccination.
  Arms: Generic Digital Intervention

SUMMARY:
The overall objective of this prospective randomized controlled study is to assess and quantify the impact of digital interventions to increase vaccination rates and vaccination-related outcomes in a connected population with self-reported diabetes. The digital intervention will be delivered via a campaign sent to participants, with interventions varying with each study arm. Participants will be blinded to study participation status.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Lives in the U.S.

Exclusion Criteria:

* < 18 years old
* Does not live in the U.S.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94321 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Evidation Health, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JL, Foschini L, Kumar S, Juusola J, Liska J, Mercer M, Tai C, Buzzetti R, Clement M, Cos X, Ji L, Kanumilli N, Kerr D, Montanya E, Muller-Wieland D, Ostenson CG, Skolnik N, Woo V, Burlet N, Greenberg M, Samson SI. Digital intervention increases influenza vaccination rates for people with diabetes in a decentralized randomized trial. NPJ Digit Med. 2021 Sep 17;4(1):138. doi: 10.1038/s41746-021-00508-2. PMID 34535755

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Existing members of the online health platform Achievement who met the inclusion criteria were blinded to their study participation status and were not asked to take any action to enroll in the study. Participants were randomized to one of the digital interventions or to no intervention. All study activities were conducted virtually.
Groups:
- People With Diabetes: Intervention: Individuals with self-reported diabetes who receive the Diabetes Digital Intervention
- People With Diabetes: Control: Individuals with self-reported diabetes who received no digital intervention
- Normal Controls-Similar: Intervention: Individuals without self-reported diabetes who were similar to PWD based on demographics and activity tracker data and received the Generic Digital Intervention
- Normal Controls-Similar: Control: Individuals without self-reported diabetes who were similar to PWD based on demographics and activity tracker data and received no digital intervention
- Normal Controls: Intervention: Individuals without self-reported diabetes and were not in NC-S based on demographics and activity tracker data, but were similar to PWD with regards to age and gender distribution and received the Generic Digital Intervention
- Normal Controls: Controls: Individuals without self-reported diabetes and were not in NC-S based on demographics and activity tracker data, but were similar to PWD with regards to age and gender distribution and received no Digital Intervention
Period: Overall Study
Arm/Group | People With Diabetes: Intervention | People With Diabetes: Control | Normal Controls-Similar: Intervention | Normal Controls-Similar: Control | Normal Controls: Intervention | Normal Controls: Controls
Started | 15702 | 15702 | 15756 | 15757 | 15702 | 15702
Completed | 5158 | 5271 | 4778 | 4810 | 5114 | 5171
Not Completed | 10544 | 10431 | 10978 | 10947 | 10588 | 10531
Not completed — Did not complete mid-study/final survey | 10544 | 10431 | 10978 | 10947 | 10588 | 10531

BASELINE CHARACTERISTICS:
Population: Overall study population
Groups:
- People With Diabetes:Intervention; People With Diabetes: Control; Normal Controls-Similar: Intervention; Normal Controls-Similar : Control; Normal Controls: Intervention; Normal Controls: Control: Participant demographics
- Total: Total of all reporting groups
Arm/Group | People With Diabetes:Intervention | People With Diabetes: Control | Normal Controls-Similar: Intervention | Normal Controls-Similar : Control | Normal Controls: Intervention | Normal Controls: Control | Total
Number analyzed (Participants) | 5158 | 5271 | 4778 | 4810 | 5114 | 5171 | 30302
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.1) | 46.7 (11.2) | 46.8 (12.4) | 46.4 (12.6) | 46.2 (12.6) | 46.6 (11.7) | 46.6 (11.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex,: Female | 4048 | 4183 | 3747 | 3814 | 4052 | 4029 | 23873
  Sex,: Male | 1096 | 1066 | 1014 | 980 | 1051 | 1128 | 6335
  Sex,: Other | 14 | 22 | 17 | 16 | 11 | 14 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3990 | 4141 | 33 | 27 | 33 | 25 | 8249
  Asian | 468 | 451 | 114 | 117 | 174 | 144 | 1468
  Native Hawaiian or Other Pacific Islander | 163 | 169 | 10 | 9 | 12 | 8 | 371
  Black or African American | 50 | 53 | 319 | 366 | 238 | 245 | 1271
  White | 19 | 18 | 3994 | 3936 | 4309 | 4453 | 16729
  More than one race | 137 | 134 | 221 | 259 | 243 | 206 | 1200
  Unknown or Not Reported | 331 | 305 | 87 | 96 | 105 | 90 | 1014
Region of Enrollment [Number; unit: participants]
  United States | 5158 | 5271 | 4778 | 4810 | 5114 | 5171 | 30302

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Self-reported Influenza Vaccination in People With Diabetes
Description: Number of participants with self-reported influenza vaccination in People With Diabetes: Intervention arm as compared to People With Diabetes: Control arm
Time Frame: 6 months
Population: 5,158 in intervention group and 5,271 in control group
Measure: Count of Participants; unit: Participants
Groups:
- Diabetes Digital Intervention: People with diabetes who received digital intervention compared to people with diabetes who did not receive digital intervention
Arm/Group | Diabetes Digital Intervention
Number analyzed (Participants) | 10429
Participants
  PWD: Intervention received influenza vaccine | 3310
  PWD: Intervention no influenza vaccine | 1848
  PWD: Control received influenza vaccine | 3220
  PWD: Control No influenza vaccine | 2051

ADVERSE EVENTS:
Time Frame: 6 months
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Groups:
- Normal Controls:Control: Individuals without self-reported diabetes and were not in NC-S based on demographics and activity tracker data, but were similar to PWD with regards to age and gender distribution and received no Digital Intervention
Arm/Group | People With Diabetes: Intervention | People With Diabetes: Control | Normal Controls-Similar: Intervention | Normal Controls-Similar: Control | Normal Controls: Intervention | Normal Controls:Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study population may not be generalizable to the entire U.S. population with diabetes. Baseline vaccination rates were relatively high and population was generally aware of their health.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT03870997/Prot_SAP_000.pdf